CLINICAL TRIAL: NCT05651919
Title: Use of Peripheral Blood Mononuclear Cells as biOmarkers of diaBetic cardIomyopathy
Brief Title: PBMC as Biomarkers of Diabetic Cardiomyopathy
Acronym: MOBI
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL22_0580; 2022-A02435-38 (Other: ID-RCB)
Record Dates: First submitted 2022-12-01; First posted 2022-12-15 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes; Metabolic Syndrome; Heart Failure With Preserved Ejection Fraction; Heart Failure With Mildly Reduced Ejection Fraction
Keywords: Type 2 diabetes; metabolic syndrome; Heart Failure with Preserved Ejection Fraction; heart failure with mildly reduced ejection fraction; PBMC
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 16 ml of blood per patient will be collected to isolate PBMC and plasma for storage at -80°C
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- No-T2D +MS / No-HF (control group): 25 patients without T2D +MS and without Heart Failure will be included in group 1.
  Interventions: Biological: Blood test; Behavioral: quality of life Questionnaire; Behavioral: Diet habits questionnaire
- No-T2D +MS / HFpEF or HFmrEF: 15 patients without T2D+MS and presenting HFpEF or HFmrEF will be included in group 2
  Interventions: Biological: Blood test; Behavioral: quality of life Questionnaire; Behavioral: Diet habits questionnaire
- T2D+MS / no-HF: 30 patients presenting T2D +MS and without any type of HF will be included in group 3.
  Interventions: Biological: Blood test; Behavioral: quality of life Questionnaire; Behavioral: Diet habits questionnaire
- T2D +MS / HFpEF or HFmrEF: 30 patients presenting T2D +MS and HFpEF or HFmrEF will be included in group 4.
  Interventions: Biological: Blood test; Behavioral: quality of life Questionnaire; Behavioral: Diet habits questionnaire

INTERVENTIONS:
Biological: Blood test — During the routine blood test of the patient, 4 more tubes of 4 milliliters (mL) will be collected to make a biological collection of PBMC and plasma for further analysis.
Behavioral: quality of life Questionnaire — During the routine medical visit, the patient will be asked to fill in a short questionnaire about quality of life.
  This is a descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems. This decision results into a 1-digit number that expresses the level selected for that dimension. Each patient's health state is referred to in terms of a 5-digit code;
  Levels of perceived problems are coded as follows:
  * Level 1 is coded as a '1' (indicating no problem)
  * Level 2 is coded as a '2' (indicating some problems)
  * Level 3 is coded as a '3' (indicating extreme problems) For example, state 11223 indicates no problems with mobility and self-care, no problems with performing usual activities, moderate pain or discomfort and extreme anxiety or depression, while state 11111 indicates no problems.
Behavioral: Diet habits questionnaire — During the routine medical visit, the patient will be asked to fill in a short questionnaire about his diet habits.
  This is an exploratory questionnaire that describes and quantifies the foods (pro- or anti-inflammatory) ingested by patients.

SUMMARY:
Type 2 diabetes (T2D), especially when associated with metabolic syndrome (MS) is at high risk to develop heart failure with preserved ejection fraction (HFpEF) or heart failure with mildly reduced ejection fraction (HFmrEF), and the specific impact of T2D+MS in cardiac function impairment is usually known as "diabetic cardiomyopathy" (DC). Cardiac remodelling (ie hypertrophy) and subtle myocardial dysfunction are highly prevalent in T2D+MS but not specific enough to predict further HFpEF or HFmrEF. Also, current biomarkers can identify but do not predict HFpEF or HFmrEF in T2D patients; Furthermore, specific biomarkers are needed. Peripheral blood mononuclear cells (PBMC) obtained from a peripheral blood sample can provide insights from calcic and inflammatory pathways, and may identify more specific molecular signatures shared between T2D+MS and HFpEF.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria common to the 4 groups:

* Patient coming for a scheduled cardiology or endocrinology visit as part of their follow-up
* Patient coming on an empty stomach for the blood test
* Male or female aged between 40 and 80 inclusive
* Patient without systemic disease and/or without anti-inflammatory treatment
* Patient not objecting to this research
* Patient accepting the conservation of biological samples and the performance of genetic analyzes

Group 1: No-T2D +MS / No-HF (control group)

* Patient without T2D or MS and without heart failure coming to a consultation or day hospital for another reason (e.g. screening for atypical symptom, etc.)

Group 2: No-T2D +MS / HFpEF or HFmrEF

* Patient without T2D or MS
* HFpEF or HFmrEF. diagnosed

Group 3: T2D+MS / no-HF

* Patient diagnosed with T2D+MS

Group 4: T2D +MS / HFpEF or HFmrEF

* Patient diagnosed with T2D and MS
* HFpEF or HFmrEF. diagnosed

Exclusion Criteria:

Non-inclusion criteria common to the 4 groups:

* History (ATCD) of cardiovascular disease (valvular (more than moderate valve disease), radiation, post-cardiotoxic chemotherapy, amyloidosis, etc.) other than HFpEF or HFmrEF
* Atrial fibrillation or permanent flutter ( paroxysmal AF is not a non-inclusion criterion: the rhythm must be sinus at the time of the ultrasound)
* Systemic disease and/or anti-inflammatory treatment
* ATCD of known coronary artery disease
* Unbalanced hypertension (>160/100 mmHg)
* Pregnant and lactating women on questioning
* Persons deprived of their liberty by a judicial or administrative decision
* Persons subject to psychiatric care
* Patients subject to a legal protection measure (guardianship, curators)
* Subject participating in another interventional research including a period of exclusion still in progress.
* Chronic kidney disease(GFR<30ml/min/1.73m2)

Group 1: No-T2D +MS / No-HF (control group)

* Presence of diabetes (whatever the type) and MS
* Presence of heart failure or other known heart disease

Group 2: No-T2D +MS / HFpEF or HFmrEF

* Presence of diabetes (whatever the type) and MS
* No Heart failure
* Left Ventricular Ejection Fraction (LVEF) on ultrasound ≤ 40%

Group 3: T2D+MS / no-HF

* Without diabetes or other type of diabetes than T2D
* Presence of Heart failure or other known coronary artery disease

Group 4: T2D +MS / HFpEF or HFmrEF

* Absence of diabetes or presence of another type of diabetes than T2D
* Absence of Heart failure
* LVEF on ultrasound ≤ 40%

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients coming at hospital for a routine visit
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-08-23 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of Initial level of Ca2+ fluxes from T2D+MS patients vs non T2D+MS patients, according to the presence or not of HFpEF or HFmrEF | Day of blood sample (inclusion visit)
  The calcic profile of PBMC will be quantified by flow cytometry to determine the values of the kinetics parameters of Ca2+ fluxes (initial level).
Comparison of amplitude of Ca2+ fluxes from T2D+MS patients vs non T2D+MS patients, according to the presence or not of HFpEF or HFmrEF | Day of blood sample (inclusion visit)
  The calcic profile of PBMC will be quantified by flow cytometry to determine the values of the kinetics parameters of Ca2+ fluxes (amplitude).
Comparison of area under curve of Ca2+ fluxes from T2D+MS patients vs non T2D+MS patients, according to the presence or not of HFpEF or HFmrEF | Day of blood sample (inclusion visit)
  The calcic profile will be quantified by flow cytometry to determine the values of the kinetics parameters of Ca2+ fluxes (area under curve).
Comparison of slope of the response to pharmacological stimulation of Ca2+ fluxes from T2D+MS patients vs non T2D+MS patients, according to the presence or not of HFpEF or HFmrEF | Day of blood sample (inclusion visit)
  The calcic profile of PBMC will be quantified by flow cytometry to determine the values of the kinetics parameters of Ca2+ fluxes (slope of the response to pharmacological stimulation).
Comparison of the inflammatory profile of PBMC from T2D+MS patients vs non T2D+MS patients, according to the presence or not of HFpEF or HFmrEF | Day of blood sample (inclusion visit)
  The inflammatory profile will evaluate by flow cytometry the proportion of the different populations of monocytes and lymphocytes using several labeling antibodies.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Louis Pradel, Bron, France